CLINICAL TRIAL: NCT06576947
Title: Effects of Virtual Reality in the Treatment of Pelvic Floor Dysfunction in Women With Multiple Sclerosis: A Randomized Clinical Trial
Brief Title: Virtual Reality in the Treatment of Pelvic Floor Dysfunction in Women With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Guadalupe Molina Torres, Senior Lecturer, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UALBIO2024/015
Record Dates: First submitted 2024-07-25; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
Keywords: virtual reality; multiple sclerosis; pelvic floor; randomized controlled trial
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind (Subject)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality therapy (Experimental): It will ve placement of virtual reality glasses that will indicate to the patient when to contract the pelvic floor.
  Interventions: Other: Virtual reality
- Neuromodulation of the tibialis posterior (Experimental): Is placed a external electrode 5 centimeters (cm) above the medial malleolus and 1 cm behind of the tibia and another electrode on the medial aspect of the foot, below the malleolus. The kind of electric current used will be rectangular, biphasic, with a pulse duration of 220 Ps and a frequency of 10 Hz. To avoid habituation to the current, a phase of 20 s stimulation with a 4 s rest phase. The intensity of the current will be inframotor, just below the contraction threshold of the flexor digitorum muscle brevis.
  Interventions: Other: Neuromodulation of the tibialis posterior nerve
- Pelvic Floor Muscle Training (Experimental): Patients will perform Pelvic Floor Muscle Training. Before performing this treatment at home, a session will be held with an expert physiotherapist in pelvic floor who will explain its implementation to the participants of this group.
  Interventions: Other: Pelvic floor muscle training

INTERVENTIONS:
Other: Virtual reality — Participants receive virtual reality treatment, 8 weeks of treatment/ 2 times a week
  Arms: Virtual reality therapy
Other: Neuromodulation of the tibialis posterior nerve — Participants receive neuromodulation of the tibialis posterior nerve8 weeks of treatment/ 2 times a week/ 30 minutes
  Arms: Neuromodulation of the tibialis posterior
Other: Pelvic floor muscle training — Participants receive pelvic floor muscle training 5 times a day for 9 weeks
  Arms: Pelvic Floor Muscle Training

SUMMARY:
The purpose of the current randomized clinical trial was to compare the effectiveness of virtual reality versus posterior tibial nerve stimulation on the improvement of pelvic floor dysfunctions in women with multiple sclerosis.

DETAILED DESCRIPTION:
* Design: Randomized Clinical Trial. Objective: to determine the effects of virtual reality versus posterior tibial nerve stimulation and muscle activation exercises on the improvement of pelvic floor dysfunctions in women with multiple sclerosis.
* Methods and Measures: forty five women will be randomly assigned to one of three groups.
* Intervention: For 8-week, the group 1 will undergo treatment with virtual reality (2/week), the group 2 will receive posterior tibial nerve stimulation (2/week) and the group 3 will receive muscle activation exercises of the pelvic floor.
* Main Outcome Measures: assessment of pelvic floor muscles function (strength and muscle tone), urodynamic studies, and validated questionnaires data will be collected at baseline, and 1 week after the last therapy application. Mixed-model analyses of variance will be used to examine the effects of the treatment on each outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Presence of pelvic floor dysfunction
* Acceptance participation
* Not undergoing another physical therapy treatment

Exclusion Criteria:

* Non-acceptance of participation
* Mental illness
* Interruption of adherence to protocolized treatment sessions
* Indication of surgical treatment in the pelvic floor

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor strength | At baseline, immediately after the intervention, and 4 weeks] [Safety Issue: No] It is a device for measuring the strength of the pelvic floor, to which a speculum is adapted. measure force in newtons
  Pelvic floor strength using a perineometer, a device for measuring the strength of the pelvic floor, to which a speculum is adapted. measure force in newtons

SECONDARY OUTCOMES:
Australian pelvic floor questionnaire: | At baseline, immediately after the intervention, and 4 weeks
  The APFQ is an instrument consisting of 42 questions in 4 domains (bladder, bowel, and sexual function and pelvic organ prolapse). relevant questions and multiplied by 10; thus, the scores range from 0 to 10 for each domain, giving a maximum total score of 40
Multiple Sclerosis Quality of Life-54 (MSQOL-54): | At baseline, immediately after the intervention, and 4 weeks
  The instrument has Likert scales and multiple-choice items. There is no single overall score for MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life). The instrument has Likert scales and multiple-choice items. There is no single overall score for MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
Euroqol | At baseline, immediately after the intervention, and 4 weeks
  It is a generic and standardized instrument developed to describe and assess health-related quality of life. The descriptive system contains five dimensions of health (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression) and each of them has three levels of severity (no problems, some problems or moderate problems, and severe problems). In this part of the questionnaire, the individual must mark the level of severity corresponding to their health status in each of the dimensions, referring to the same day they completed the questionnaire. In each dimension of the EQ-5D, severity levels are coded as 1 if the response option is "I have no problems"; with a 2 if the response option is "some or moderate problems"; and with a 3 if the answer option is "many problems." The higher score meaning a worse result.
SF12 | At baseline, immediately after the intervention, and 4 weeks
  This questionnaire contains 12 items that assess 8 aspects of HRQoL: physical dimension, mental dimension, physical function, physical role, bodily pain, general health, vitality, emotional role, social function, and mental health. The SF-12 v2 response options form Likert-type scales that evaluate intensity or frequency. The number of response options ranges between three and six, depending on the item, and each question receives a value that is subsequently transformed into a scale from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Molina Torres, Principal Investigator — Universidad de Almeria; Jacobo Ángel Rubio-Arias, Principal Investigator — Universidad de Almeria; Marta María Córdoba Peláez, Principal Investigator — Universidad de Almeria